CLINICAL TRIAL: NCT07366229
Title: Evaluating Engineered Lactobacillus Reuteri With a Zinc Sulfate-Tannic Acid MPN Coating for Acne: A Double-Blind, Randomized Controlled Trial
Brief Title: Topical Application of Engineered Lactobacillus Reuteri With a Zinc Sulfate-Tannic Acid MPN Coating for Acne
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LL-KY-2025172-02
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Acne
Keywords: acne; Lactobacillus reuteri
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Experimental Group Intervention: Apply the MPN-coated engineered Lactobacillus reuteri cream to acne lesions once daily for 2 weeks.
  Control Group Intervention: Apply the plain Lactobacillus reuteri cream to acne lesions once daily for 2 weeks.
  Negative Control Group Intervention: Apply the petrolatum-glycerin cream to acne lesions once daily for 2 weeks.
  Positive Control Group Intervention: Apply the 0.1% tretinoin cream to acne lesions once daily for 2 weeks.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group (Experimental): Apply the MPN-coated engineered Lactobacillus reuteri cream to acne lesions once daily for 2 weeks.
  Interventions: Biological: MPN-coated engineered Lactobacillus reuteri cream
- Positive Control Group (Active Comparator): Apply the 0.1% tretinoin cream to acne lesions once daily for 2 weeks.
  Interventions: Drug: Tretinoin cream 0.1%
- Negative Control Group (Placebo Comparator): Apply the petrolatum-glycerin cream to acne lesions once daily for 2 weeks.
  Interventions: Drug: Petrolatum-glycerin cream
- Control Group (Other): Apply the plain Lactobacillus reuteri cream to acne lesions once daily for 2 weeks.
  Interventions: Biological: Plain Lactobacillus reuteri cream

INTERVENTIONS:
Biological: MPN-coated engineered Lactobacillus reuteri cream — Each night before bedtime, after washing the face, an appropriate amount of MPN-coated engineered Lactobacillus reuteri cream should be applied topically to acne lesions using a sterile cotton swab. The area should not be washed immediately after application. Normal face washing can be resumed the following morning. This regimen should be continued for 2 weeks.
  Arms: Experimental Group
Biological: Plain Lactobacillus reuteri cream — Each night before bedtime, after washing the face, an appropriate amount of plain Lactobacillus reuteri cream should be applied topically to acne lesions using a sterile cotton swab. The area should not be washed immediately after application. Normal face washing can be resumed the following morning. This regimen should be continued for 2 weeks.
  Arms: Control Group
Drug: Petrolatum-glycerin cream — Each night before bedtime, after washing the face, an appropriate amount of petrolatum-glycerin cream should be applied topically to acne lesions using a sterile cotton swab. The area should not be washed immediately after application. Normal face washing can be resumed the following morning. This regimen should be continued for 2 weeks.
  Arms: Negative Control Group
Drug: Tretinoin cream 0.1% — Each night before bedtime, after washing the face, an appropriate amount of 0.1% tretinoin cream should be applied topically to acne lesions using a sterile cotton swab. The area should not be washed immediately after application. Normal face washing can be resumed the following morning. This regimen should be continued for 2 weeks.
  Arms: Positive Control Group

SUMMARY:
A growing body of evidence suggests that the development and progression of acne are closely linked to an imbalance in the skin's microbial community. Compared to healthy skin, the composition and function of the microbiota in acne lesions are significantly altered. This microbial imbalance is believed to drive the formation and recurrence of acne through mechanisms such as triggering abnormal inflammatory responses and compromising the skin barrier.

An in-depth exploration of the interaction between acne and the skin microbiome not only offers new perspectives for understanding the root causes of the disease but also lays the groundwork for developing novel treatment strategies aimed at modulating the microbiota. Therefore, identifying innovative approaches that integrate acne treatment with the regulation of microbial balance holds significant clinical and social value.

Although existing acne treatments have made progress, research focusing on interventions that regulate the local skin microecology through probiotics remains relatively limited. This study aims to explore a new strategy based on skin microecological modulation. We are using a common probiotic-Lactobacillus reuteri-and applying an engineering modification with a special coating formed by zinc sulfate and tannic acid (MPN coating). This modification is intended to enhance the bacterium's survival and colonization on the skin, thereby more effectively regulating the local microbiota and reducing inflammation.

This study is a rigorous scientific clinical trial designed as randomized, double-blind, and controlled. Eligible participants will be randomly assigned to one of four groups, receiving either the engineered Lactobacillus reuteri cream, the plain Lactobacillus reuteri cream, a simple moisturizing cream (placebo), or an already-marketed effective cream (tretinoin cream). The treatment will last for 2 weeks, followed by an 8-week observation period. Efficacy and safety will be evaluated through professional assessments.

Our goal is to scientifically evaluate the safety and efficacy of this new therapy, hoping to provide a potential new treatment option for individuals with acne and explore new pathways for improving skin health.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be diagnosed with acne (based on history, clinical manifestation, and dermatoscopy) and classified as Grade I to III per the International Improved Grading System.
2. Subjects must be willing and able to provide written informed consent.
3. Subjects must be 18 to 33 years of age and in generally good health.
4. Subjects must have more than 9 inflammatory lesions.

Exclusion Criteria:

1. Have used antibiotics within 1 month before the study start.
2. Have used systemic retinoid therapy within 3 months before the study start.
3. Have undergone any other acne treatment within 1 month before the study start.
4. Have any other condition that the investigator considers would make participation unsuitable (e.g., deemed unreliable, non-compliant, or unable to comprehend the study assessments).

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage change in acne count at Week 8 relative to the baseline. | Facial photographs of the patients will be taken at baseline and at Weeks 1, 2, 4, and 8 after the initial treatment, and the number of acne lesions will be counted by dermatologists.
  Facial photographs of patients are taken before treatment and at Weeks 1, 2, 4, and 8 after the initial treatment. Dermatologists count the number of acne lesions from these photographs. The percentage change in acne count at Week 8 relative to the baseline is calculated as: (Acne count at Week 8 - Acne count at baseline) / Acne count at baseline × 100%.

SECONDARY OUTCOMES:
Percentage change in the number of inflammatory acne lesions at Week 8 relative to the baseline | Facial photographs of the patients will be taken at baseline and at Weeks 1, 2, 4, and 8 after the initial treatment, and the number of inflammatory acne lesions will be counted by dermatologists.
  Facial photographs of patients are taken before treatment and at Weeks 1, 2, 4, and 8 after the initial treatment. Dermatologists count the number of inflammatory acne lesions from these photographs. The percentage change in the number of inflammatory acne lesions at Week 8 relative to the baseline is calculated as: (Number of inflammatory acne lesions at Week 8 - Number of inflammatory acne lesions at baseline) / Number of inflammatory acne lesions at baseline × 100%.
Percentage change in the number of non-inflammatory acne lesions at Week 8 relative to the baseline | Facial photographs of the patients will be taken at baseline and at Weeks 1, 2, 4, and 8 after the initial treatment, and the number of non-inflammatory acne lesions will be counted by dermatologists.
  Facial photographs of patients are taken before treatment and at Weeks 1, 2, 4, and 8 after the initial treatment. Dermatologists count the number of non-inflammatory acne lesions from these photographs. The percentage change in the number of non-inflammatory acne lesions at Week 8 relative to the baseline is calculated as: (Number of non-inflammatory acne lesions at Week 8 - Number of non-inflammatory acne lesions at baseline) / Number of non-inflammatory acne lesions at baseline × 100%.
Changes in the relative abundance of Propionibacterium, Lactobacillus, and Staphylococcus in acne-prone skin from baseline to Week 8 | Skin microbiome samples are collected from acne lesions at baseline and at Weeks 1, 2, 4, and 8 after the initial treatment.
  Skin microbiome samples are collected from acne lesions before treatment and at Weeks 1, 2, 4, and 8 after the initial treatment. These samples are subjected to 16S rRNA gene sequencing to detect the presence and relative abundance of various bacterial taxa in the affected areas following the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No